CLINICAL TRIAL: NCT06523686
Title: Lateral Ridge Augmentation Using Autogenous-xenogeneic or Allogeneic-xenogeneic Graft Mix With a Cross-linked Collagen Membrane: a Randomized Pilot Clinical Trial
Brief Title: Lateral Ridge Augmentation Using Two Graft Combination and a Cross-linked Collagen Membrane
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Celine Rassi, Periodontology resident, Saint-Joseph University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USJ-2023-57
Record Dates: First submitted 2024-07-10; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Alveolar Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogeneic-xenogeneic combination (Experimental): A mix of 2/3 allogeneic bone with 1/3 xenogeneic bone
  Interventions: Procedure: Guided bone regeneration
- Autogenous-xenogeneic combination (Experimental): A mix of 2/3 autogenous bone and 1/3 xenogeneic bone
  Interventions: Procedure: Guided bone regeneration

INTERVENTIONS:
Procedure: Guided bone regeneration — Compare the linear and volumetric bone width changes, clinically and radiographically, between two different bone graft combinations (autogenous-xenogeneic and allogeneic-xenogeneic) covered with a cross-linked collagen membrane in a horizontal GBR.

SUMMARY:
To treat resorbed alveolar ridges, many surgical procedures are available in the literature such as ridge splitting, distraction osteogenesis, block grafting techniques and guided bone regeneration, which is the most documented technique. Various grafting materials are available but there is a lack of evidence on the superiority of a material or a combination of materials.

DETAILED DESCRIPTION:
Bone width at the implant site is an important prerequisite for a predictable and long-term prognosis in implant dentistry. Different types of membranes and bone grafts are used in the GBR procedure. However, there is a lack of studies in the literature about the combination allograft/xenograft. The aim of the present trial is to compare two different bone graft combinations (autogenous-xenogeneic and allogeneic-xenogeneic) covered with a cross-linked collagen membrane in a horizontal alveolar ridge augmentation (without simultaneous implant placement).

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, non-smokers or smokers <10 cigarettes/day.
* Age between 20 and 75.
* Full mouth bleeding score (FmBS) <20 %.
* Full mouth plaque score (FmPS) <15%.
* Residual bone width < 5 mm and adequate bone height in the maxilla and the mandible.
* Tooth extraction performed at least 6 weeks before surgery.
* Presence of enough teeth to support an occlusal stent/radiographic guide.

Exclusion Criteria:

* Systemic diseases.
* Heavy smokers (> 10 cigarettes/day).
* History of radiotherapy in the head and neck region in the last 5 years.
* Active periodontitis on the remaining teeth.
* Pregnancy.
* Intake of medications that may have an effect on bone turnover and mucosal healing (i.e., tetracycline within the last month, steroids within the last 6 months, bisphosphonates or fluorides at bone therapeutic levels, vitamin D and metabolites at therapeutic levels within the last 6 months).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Linear bone width changes | 6 months
  Linear bone width changes assessed clinically and radiographically in mm
Volumetric bone changes | 6 months
  Volumetric bone changes assessed radiographically in cubic mm

SECONDARY OUTCOMES:
Clinical Ridge Height gain | 6 months
  Clinical Ridge Height gain in mm
Probe penetration | 6 months
  Probe penetration at the occlusion-buccal angle

CONTACTS AND LOCATIONS:
Overall Officials: Celine Rassi, DDS, Principal Investigator — Saint-Joseph University
Locations (1):
- Saint Joseph university, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No